CLINICAL TRIAL: NCT00155636
Title: A Study on Etiological Factors of Schizophrenia
Status: Terminated | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 5287; NHRI-EX91-9113PP
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2002-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This PPG entitled "A Study on Etiological Factors of Schizophrenia" (SEFOS) focuses on searching for the separate etiological factors under the understanding that schizophrenia is a complex disorder. Multifactorial model has been most often proposed as the etiological model. Up to now, fragmented knowledge of etiological factors, including genetic factor and environmental insults were reported in literature, and a two-strike hypothesis has been proposed. This PPG of SEFOS formulates a dynamic etiological hypothesis of schizophrenia. Specific, however heterogeneous, genes are hypothesized to be located in chromosome 1q, 6P, 8P, 15q, and 22q; specific environmental insults or stress are hypothesized to be acting in the vulnerable brain a long different stages of biological and/or psychological development. The interaction of specific genes and specific environment insults/stress along different stages of development will result in specific neurobiological abnormalities as shown in neuropsychological, neurophysiological and neurochemical/neuroimaging abnormalities. For this hypothesis testing, this PPG of SEFOS designs 3 projects of: (1) A Study on Neurobiology of Schizophrenia; (2) A Study on Environmental insults/stress of schizophrenia; and (3) Molecular Genetics Study of Schizophrenia. Project No.1 aims at finding different levels of neurobiological and anatomical abnormalities; Project No.2 aims at finding different levels of environmental insults/ stress; Project No.3 aims at locating vulnerability genes in different chromosome regions. A core unit for administrative integration, for case/family recruitment and statistical analysis is also designed. The dynamic etiological complex will be explored under multivariate statistical analysis. This PPG of SEFOS adopts multidisciplinary approach including clinical psychiatrists, psychopathologists, neuropsychologist, neurophysiologist, neuroimaging (magnetic resonance imaging) specialist, genetic epidemiologist, molecular genetic specialist, genetic statistician, and biostatisticians. This team has sound mutual trust base on the experience of being working together and attending regular research meeting for the part several years under the leadership of the principal investigator of this PPG.

DETAILED DESCRIPTION:
Progress Report Schizophrenia is a chronic and devastating major psychiatric disorder. It costs a lot of the individual patient, the family as well as the society. Schizophrenic patients occupy around 80% of the chronic psychiatric beds. About 60 % of the acute psychiatric beds serve the schizophrenic patients at severe aggravating state of illness. The majority of the schizophrenic patients need the support of the family for their daily life. For better service of these patients, their family as well as for reducing social stigma of schizophrenia patients, more psychopathological understanding is crucial. However, schizophrenia is a complex disorder. For the past one century, the understanding of schizophrenia improved much. In Taiwan, the psychopathological study on schizophrenia deserves basic and systematic approach for clinical and academic purpose.

Before it could be possible to understand the essence of the psychopathology of schizophrenia, the descriptive psychopathology has to be well documented. The heterogeneity at the level of clinical pathology has to be delineated as the initial step of psychopathological study of schizophrenia. This is crucial under the consideration of cross-cultural application of diagnostic criteria in the definition of schizophrenia. The psychopathology of the disease category of schizophrenia as defined by the DSM-IV system was documented mainly by the literature based on the descriptive study of the patients of the Caucasian population and the related culture. Western medicine in Taiwan is totally accepted in the academic circle. From a cross-cultural point of view, this way of academic operation has to be reflected methodologically and to be examined empirically.

Research on schizophrenia psychopathology has to be of two kinds of value. The first is to be of the frontier academic work of the World Psychiatry, and the study results can contribute to the knowledge of the World Psychiatry Literature. The second is to be of native cultural value. The results could be of value in reflecting the native cultural reality and could be of value in application of these study results to clinical service.

To be at the frontier of schizophrenia research, the neuropsychological impairments underlined the clinical manifestations of schizophrenia is one major area of study. In contrast to the traditional theory of psychological defense mechanism or the psychosocial explanation of psychopathology of schizophrenia, the neuropsychological approach could provide the way to understand the neural mechanism of schizophrenia psychopathology at the level of psychological function. In the era of neuroscience achievement, this approach is promising and crucial.

The most basic psychopathology of schizophrenia is the genetic factor of etiology. In the era of molecular medicine, the genetic epidemiological and molecular genetic study on schizophrenia psychopathology is the most frontier line of schizophrenia research.

This research team leaded by the Principal Investigator, Hai-Gwo Hwu, of this PPG began this approach in July 1993. The initial work started with the Multidimensional Psychopathological Group Research Project: Schizophrenia" (MPGRP). This MPGRP was designed based on the theoretical evolutionary model (EM) of psychopathology invented by this Principal Investigator. This EM model included multiple psychopathological factors including genetic factors, brain insults, chronic developmental life experience, neurobiological manifestations, personality-adjustment factor, environmental stress of biological and psychological factors, familial social cultural value factor and the factor of treatment. In this EM model, the disease course was hypothesized into three phases: initial subclinical stage, clinical stage, and the outcome stage after treatment. This MPGRP was thus designed following the guidance of EM psychopathological model.

To design the psychopathological study based on this EM of psychopathology, it is necessary to invent a new methodological approach. This approach included serial multi-dimensional study design. The first step was to set-up a smooth infrastructure and to collect a cohort of clinical schizophrenia cases for follow-up study, and also to collect schizophrenia family with at least two siblings affected with schizophrenia for molecular genetic study. This first step also considered that the descriptive psychopathological study, the study on search for a biological trait marker and the search for identification of linkage of possible vulnerability genetic markers of schizophrenia as the major research tasks.

The initial project started as the MPGRP from July 1993 till June 1998, the subsequent project following the initial MPGRP, was the Multidimensional Psychopathological Study on Schizophrenia (MPSS) started in July 1998 till June 2001. The focus of the MPGRP was to study the clinical manifestations of schizophrenia and the family situation in a cohort of schizophrenia patients. The MPGRP also focused on the phenotype definition of schizophrenia using CPT manifestation in the schizophrenia family. CPT was done in all of the family of schizophrenic patients. The family with at least two siblings affected with schizophrenia were collected for molecular genetic study.

In the MPSS project, the focus was on the follow-up neuropsychological evaluation of the schizophrenia cohort collected in the MPGRP, other than the descriptive follow-up clinical data collection. Besides, the MPSS also focus on the CPT and WCST studies on the family members o the family with at last two siblings affected with schizophrenia. These families are also the sample for molecular genetic study. The collection of the schizophrenia family of this kind for molecular genetic study is still the work of this MPSS, as the collection of this kind of family was not an easy task.

There are several important features characterize the uniqueness of this MPGRP and MPSS : (1) a prospective follow-up design, (2) multidisciplinary approach, (3) multi-center, multi-hospital approach, (4) operationalized assessment of schizophrenia psychopathology using the "Positive and Negative Syndrome Scale" (PANSS)(4), (5) covering multi-dimensional psychopathological factors, (6) representing up-to-date psychopathological study of phenotype definition, molecular genetic study, neuropsychological study, as well as the study on the expressed emotion of the chief care giver and the family burden and need of care of the patients.

This MPGRP and the MPSS were successfully carried out from July 1993 to March 2001(up to the time of sending this SEFOS proposal as the subsequent study on the pathogenesis of schizophrenia, a further step of psychopathological study on schizophrenia) based on the following facts:

1. This MPGRP and the MPSS made the multidisciplinary team to be possible in psychopathological study in Taiwan. This is not an easy task. Other than the technological breakthrough in research administration in this manner, the successful element was that this multidisciplinary approach made a smooth working infrastructure for this psychopathological research for successive research works. Other than research work itself, the attending members of this research team obtained continuous training and exercise in psychopathological study. These achievements cannot be demonstrated in literature publication.

2. This MPGRP and the MPSS made the multi-center, multi-hospital approach came true in Taiwan in psychopathological study. This institutional infrastructure guarantee that the sampling of schizophrenic cases to be more representative of patient population for psychopathological study. Other than research administration breakthrough, this approach provided a great chance for clinical psychiatrist to participate in training and practice in psychopathological basic training. Besides, the clinical service team members, other than psychiatrist, including psychiatric nurse, psychologist, psychiatric social worker can obtain the common sense understanding of general psychopathological approach in psychiatry. This close team approach will make the service team to be more cohesive in the care of the patients. The patients attending this study would obtain more attention from the psychiatric service team leaded by the research psychiatrist, especially in the successive follow-up study. This is crucial in elevating the professional activity in a positive sense embedded in this MPGRP and MPSS research. This is also one achievement of this MPGRP and MPSS in the infrastructure of this research approach. These achievements cannot be demonstrated in literature publication, but can be demonstrated in daily research and practice activities. It can also be shown in the subsequent research activities such as this SEFOS project.

3. This MPRP and MPSS brought the Taiwan Psychiatry to the frontier line of psychopathological study and contribute new knowledge to schizophrenia literature. Besides, this MPGRP and MPSS also took care of the standpoint of the native culture background. The descriptive phenomenological approach is the essence of operationalized psychopathological study. The cross-cultural modification and justification of the Western rating schedule of the PANSS has been considered and successfully done.

4. The family of schizophrenic patent was also the major area of study based on the characteristics of the Taiwan culture. The family took the responsibility of patient care closely. The burden and the need of patient care are important topic of this study. Besides, taking the advantage of the culture background of the close family tie of the patient and the family, genetic study of schizophrenia including genetic epidemiology and molecular genetics is one major task of this MGRP and the MPSS too.

5. Major academic achievements of the track of this PPG and the MPSS psychopathological study in these past 7 to 8 years included the following:

1. The findings of different symptom clusters of schizophrenia:

   Categorical or dimensional approach of schizophrenia psychopathology is still a current unsolved issue in schizophrenia research. The MPGRP collected 234 schizophrenia subjects in the Northern part of Taiwan and designed a cohort follow-up study in 1993. At the end of this MPGRP, ranged from1998 to 2000 for data analysis, the descriptive psychopathological PANSS data assessed on admission were analyzed using explorative factor analysis (EFA) and confirmatory factor analysis (CFA), and a basic 4- dimensional model of schizophrenia psychopathology was established. These 4 dimensions are: "Negative and associated Negative symptoms", "Disorganized thought", "Hostility/excitement", and "Delusion/hallucination". Including the general psychopathological section of the PANSS, there is an additional dimension of anxiety/depression was found in the EFA. The CFA cannot found satisfactorily model for model fitting as the general psychopathology section was included in CFA. This could be due to the high variability and low base rates of these items of the general psychopathological section of PANSS. Besides, this could also be due to the peripheral nature of these symptom items in schizophrenia psychopathology.

   These findings were confirmed by another statistical graphic approach, the color graphic generalized association plots (GAP) in delineating the heterogeneity of descriptive symptom pathology of the schizophrenia. In this GAP analysis, again a 4-dimension model was also found based on the PANSS data assessed on admission. These 4 dimensions were also arranged according to the proximity matrix and were revealed as the following order: (1) "Negative symptom", (2) "Disorganized thought", (3) "Hostility/Excitement". (4) "Delusion/hallucination" dimensions. The possible dimension of "Anxiety/depression" was also observed near the end of the dimension of "Negative symptom dimension".

   The validity of these symptom dimensions was assessed using the impairment of sustained attention assessed by continuous performance test (CPT). It was found that the negative symptom dimension was associated with impaired CPT. Furthermore, the severely impaired (Z>3.0) d' of CPT was found to be associated with persistent negative symptom, the deficit state of clinical psychopathology, of schizophrenia. The delusion/hallucination dimension was found to be associated with the impaired neuronal activity of hippocampal region measured by the neuroimaging technology of Magnetic Resonance Spectrometry (MRS).

   The GAP analysis based on the successive PANSS data assessed on admission, 6-month, 1-year and 2-year follow-up also showed a stable 5-dimension model of psychopathology. The component symptom dimensions were the same as that of the data assesses on admission. These are dimensions of "Negative symptom", "Disorganized thought", "Hostility/excitement", "Delusion/hallucination" and "Anxiety/depression". This research team developed the concept of core symptom dimension by selecting the stable symptom items appeared stably over the all follow up course over 4 successive assessments across the 2-year follow-up. The validity of these core psychopathological dimensions composed of core, stable symptom cluster items is still under investigation.
2. The findings of different subgroups of schizophrenia patients:

   Based on the cohort follow-up design, it is possible to search the possibility of the existence of different subgroups of patients be categorical approach. Matched with the effort on differentiating the symptom dimensions of psychopathology, it is also possible to define the different subgroups of patients based on the composition of symptom dimensions. This research team invented this analytical approach called as the GAP analysis for this purpose. The results were partly shown in the website: http://gap.stat.sinica.edu.tw. Based on the admission PANSS data, this GAP found 4 symptom clusters of "Negative symptom", "Disorganized thought", "Hostility/excitement", and "Delusion/hallucination", and also two subgroups of patients with (GWNEG) and without (GONEG) marked negative symptoms. These two groups of patients were found to have validity from the manifestation of clinical symptom dimensions in the follow-up course and CPT performance. Besides, these two subgroups also differed in the treatment response an prognostic outcome as shown in social functions.

   The GAP analysis, based on the follow-up data of PANSS assessment, can also find consistently a 4 -dimensional model of schizophrenia psychopathology. One additional dimension of anxiety/depression was also found. The patient subgrouping consistently found three patient subgroups at 6-month, 1-year and 2-year follow-up. One is of low psychopathology group (good treatment response group), the other is of marked blunt group and the last is of persistent delusion/hallucination group. The concordance of the GWNEG and GONEG and these three groups are still under investigation.
3. Impaired sustained attention by continuous performance test (CPT) as the trait marker of schizophrenia.

   We used a CPT machine from Sunrise Systems, version 2.20 (Pembroke, MA, USA). The procedure has been described in detail I our publications. Briefly, numbers from 0 to 9 were randomly presented for 50 milliseconds each, at a rate of one per second. Each subject undertook two CPT sessions: the undegraded 1-9 task and the degraded 1-9 task. The sensitivity index (d) of the CPT performance reflects the subject's sustained attention. Family studies have indicated that sustained attention deficits as measured by the CPT are vulnerability markers of schizophrenia. The results are: (1) a substantial proportion of non-psychotic relatives of schizophrenia probands (19-34%) have CPT deficits, which can be predicted from their probands' CPT performance; (2) subjects with schizotypal personality features also exhibit CPT deficits, which are specifically associated with negative factors of schizotypy; (3) CPT deficits are present in schizophrenic patients, are particularly associated with negative and disorganized symptoms, and those with more difficult CPT versions are not amenable to neuroleptic treatment.
4. The familial tendency of schizophrenia in Taiwan schizophrenia proband In this MPGRP and MPSS stdy, the Diagnostic Interview Schedule for Genetic Study (DIGS) and schizotypy interview schedule (SIS) were translated and modified to be useful in Taiwan subjects. The Perceptual aberration scale (PAS) and Schizotypal personality questionnaire (SPQ) were also used in community study on schizophrenia-related personality disorders. The cross-cultural consideration was employed. In community study, the schizophrenia-related personality disorders were assessed using the PAS and SPQ initially and then by DIGS and SIS interview. Including schizophrenia-related personality disorder in the spectrum did not increase power for linkage analysis o schizophrenia. This is one important information for our molecular genetic study of this MPGRP and MPSS.
5. Explorative neurobiological study on the schizophrenic samples of this MPGRP and the MPSS project.

   The neuropsychological study of the MPSS design and the impact of the concept of endophenotype of molecular genetic study induce this MPSS research team to explore the role of the neurophysiological parameter of P50 inhibition and the neurochemical parameter of neuronal activity shown in Magnetic Resonance Imaging Spectrometry (MRS) of relative concentrations of various specific biochemical molecules such as choline and creatinine.

   The P50 study and the related neurophysiological study provided the chance to study the implicit and explicit study paradigm of schizophrenia. The implicit learning of color in schizophrenia was fond to be significantly impaired as compared to the controls. The 3-D dimension display of brain energy in this P50 study showed that the energy distribution of the schizophrenic patients was significantly different from that of the controls. The MRS study showed that the positive symptom cluster was correlated to the decreased neuronal activity of the hippocampal region. These study results make it possible for this research tem to design the research on the all family members of the schizophrenia proband for pathogenesis genetic study on multi-etiological factors and their interaction by using these neurobiological parameters designed in this SEFOS, an investigation on the dynamic pathogenetic process of schizophrenia, leaded by this Principal Investigator with smooth working infrastructure for multidimensional psychopathological study on schizophrenia.
6. Molecular genetic study on locating vulnerability gene in different chromosome regions.

   Linkage study and association study were performed in this project for locating the vulnerability genes of schizophrenia by examining the warm spots of schizophrenia in some chromosome regions of chromosome 1q, 6p, 8p, and 15q. The study results, so far obtained in this laboratory using 52 Taiwanese families with at least 2 siblings affected with schizophrenia, could not exclude the possible existence of the schizophrenia vulnerability genes locations in these chromosome regions.

   Further study of the PPG of SEFOS will focus on these positions of these 5 markers with potential linkage to find closer genetic markers possibly linked with schizophrenia using closer genetic markers such as the combination of dinucleotide and SNP markers. The candidate genes around these genetic markers will also be explored to search for mutations related to the pathological variation of schizophrenia. This will be the focus of this PPG of SEFOS too following this MPGRP and MPSS.

   This laboratory is exploring for the possibility of the candidate gene approach based on plausible animal model of schizophrenia and/or pathophysiological process of schizophrenia. The NMDA subunit R1 receptor gene and nicotinic receptor alpha 7 subtype genes are two genes under exploration. The skin test of niacin test was also explored in this laboratory for the possible association with genetic defect in the phospholipid metabolism related genes. These will be included in this PPG of SEFOS study in the future.
7. Expressed emotion and burden of the family of schizophrenic patients The family as a unit of study is also concerned in this MPGRP and the MPSS. The expressed emotion was once considered to be a stable trait of the family chief caregiver and was hypothesized to have specific psychopathological meaning in schizophrenia. However, the expressed emotion of the Taiwanese schizophrenia family was found to be changing according the course of illness. It was not stable. The family burden was found to be very high and specific clinical measures for relieving thee family burden has to be designed for better clinical service of the schizophrenia family.
8. Invention of statistical method for psychopathological study The multivariate nature of the psychopathological data demands the invention of novel statistical method for data management. In this MPGRP and the MPSS, the analysis of 33 PANSS symptoms and the subgrouping of the patients in the study of schizophrenia heterogeneity invite a development of the new color graphic approach in the exploration of symptom dimensions and patent subgrouping. This was named as Generalized Association Plots (GAP). This demonstrates the fruitful approach in the multi-disciplinary team-work in the psychopathological study.
9. Data bank establishment of this MPGRP and the MPSS. In the past 7 to 8 years of the MPGRP and MPSS work, important data banks of clinical psychopathology of schizophrenia were established. These data banks will be useful for successive data analysis to test the various hypotheses related to the issues of heterogeneity of schizophrenia. These data banks included (1) basic clinical data bank of schizophrenia cohort of 234 cases and their follow-up clinical data for up to 7 years of follow-up data, (2) data bank of objective ratings of PANSS, ESRS, and CDRS, and (3) neuropsychological testing data bank of successive follow-up neuropsychological evaluations. The DNA bank and cell-line bank of the families of schizophrenia and other related disorders is also very important for further molecular genetic evaluation.

Other than this DNA data bank of this MPGRP and MPSS, this laboratory also performed the Taiwan Schizophrenia Linkage Study (TSLS) in collaboration with researchers of the Harvard Medical School under the support of the NIMH, U.S.A., to collect 600 families with at least two siblings affected with schizophrenia. This data bank included DIGS, DNA and CPT as well as WCST. This research team will use this data set to replicate the initial findings obtained in this laboratory originally. This will be one major focus of the subsequent SEFOS of this PPG.

All these data banks justify the abundant resource of data for continuous data analysis and paper publication of this SEFOS of the PPG, and this is the reason that this SEFOS has to set the core containing a statistical sub-core unit for the operation of data analysis. Up to the present, this research team is mature enough to do continuous data analysis and serial hypothesis testing. All these data provided the evidence that the grant of this SEFOS will, apparently, achieve the expected results of this research team with great confidence.

6. The progress of the MPSS (July, 1998 - June 2001) till March, 2001 as the PPG of SEFOS was proposed. Three sub-projects were reported to be as the following:

1) Phenomenological and neuropsychological manifestations of schizophrenia: a prospective follow-up study.

(2) A family-genetic study of co-affected sib-pairs with schizophrenia. (3) Molecular genetic study on schizophrenia using co-affected sib-pair and association strategies.

In conclusion, this MPSS has been going on smoothly in data collection as well as in data analysis. The paper publication is going on steadily. These three sub-projects were integrated and coordinated smoothly. Besides, the preliminary works using the neurobiological technology of neurophysiology and brain Magnetic Resonance Spectrometry (MRS) for measurements of psychopathological related manifestations have been performed. These technologies were proved to be satisfactorily stable and applicable in psychopathological study. The preliminary results were obtained and manuscripts were prepared for submission. Actually, the technology can also be extended to the other brain parts including the frontal region and the measurement of tractography is also available in the imaging laboratory of the National Taiwan University Hospital.

The past tract record of the achievement of the smooth working infrastructure of this research team leaded by the P.I. Hai-Gwo Hwu, including multidisciplinary specialists and multi-institutes, the achievement of the advanced technologies of neurobiological measurements related to the study of current psychopathological investigation of schizophrenia, the previous achievement in psychopathological hypothesis testing and the academic achievement of this research team, and the abundant data bank, highly justify that this research team of the SEFOS of this PPG is a well cultivated research tem in schizophrenia research. This SEFOS of PPG can positively be expected to have successful results in the future if this team has this SEFOS grant for the coming 5 years of research work.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* There are two schizophrenia sib-paired children, one schizophrenia parent and the other one should be normal

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1056
Dates: Start 2002-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Gwo Hwu, Professor, Principal Investigator — National Taiwan University